CLINICAL TRIAL: NCT02474498
Title: Enamel Matrix Protein Derivative and/or Synthetic Bone Substitute for the Treatment of Mandibular Class II Buccal Furcation Defects. A 12-month Randomized Clinical Trial
Brief Title: EMD and/or Bone Substitute for the Treatment of Class II Furcations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Professor, department of Periodontics, Piracicaba Dental School, State University of Campinas (UNICAMP), Piracicaba, São Paulo, Brazil, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 035/2007
Record Dates: First submitted 2015-06-10; First posted 2015-06-17 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2015-06

CONDITIONS: Periodontal Disease
Keywords: Regenerative therapy; Randomized clinical trial (RCT); Enamel matrix derivative; Hydroxyapatite-beta tricalcium phosphate; Buccal furcation
MeSH Terms: conditions — Periodontal Diseases | interventions — enamel matrix proteins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EMD alone (Active Comparator): During flap access surgery, the granulation tissue will be removed and the root surfaces will be carefully instrumented with ultrasonic and hand instruments. The furcation defects in this group will receive the application of enamel matrix derivative (EMD - Emdogain® Straumann, Basel, Switzerland) and after the flap will be repositioned.
  Interventions: Drug: EMD; Procedure: Flap access surgery
- βTCP/HA alone (Active Comparator): During flap access surgery, the granulation tissue will be removed and the root surfaces will be carefully instrumented with ultrasonic and hand instruments. The furcation will be filled with a bone substitute consisting of beta tricalcium phosphate/hydroxyapatite (βTCP/HA- Bone Ceramic® Straumann, Basel, Switzerland)
  Interventions: Device: βTCP/HA; Procedure: Flap access surgery
- EMD + βTCP/HA (Active Comparator): During flap access surgery, the granulation tissue will be removed and the root surfaces will be carefully instrumented with ultrasonic and hand instruments. The furcation will be filled with a mixture of enamel matrix derivative proteins (EMD) (Emdogain® Straumann, Basel, Switzerland) and bone substitute consisting of βTCP/HA (Bone Ceramic® Straumann, Basel, Switzerland). Immediately after debridement, EMD will be applied on the root surfaces. The remaining part of the material in the seringe will be then mixed with the bone substitute on a sterile dappen. This mixture will be used to completely fill the defect (EMD + βTCP/HA).
  Interventions: Drug: EMD; Device: βTCP/HA; Procedure: Flap access surgery

INTERVENTIONS:
Drug: EMD — During flap access surgery, the granulation tissue will be removed and the root surfaces will be carefully instrumented with ultrasonic and hand instruments. The furcation defects in this group will receive the application of enamel matrix derivative (EMD - Emdogain® Straumann, Basel, Switzerland).
  Other Names: Emdogain
  Arms: EMD + βTCP/HA; EMD alone
Device: βTCP/HA — During flap access surgery, the granulation tissue will be removed and the root surfaces were carefully instrumented with ultrasonic and hand instruments. The furcation will be filled with a bone substitute consisting of beta tricalcium phosphate/hydroxyapatite (βTCP/HA- Bone Ceramic® Straumann, Basel, Switzerland)
  Other Names: Bone Ceramic®
  Arms: EMD + βTCP/HA; βTCP/HA alone
Procedure: Flap access surgery — In the furcation sites, during flap access surgery, the granulation tissue will be removed and the root surfaces will be carefully instrumented with ultrasonic and hand instruments.

SUMMARY:
To clinically evaluate the treatment of mandibular class II furcation defects with enamel matrix derivative (EMD) and/or a bone substitute graft make of beta tricalcium phosphate/hydroxyapatite (βTCP/HA).

DETAILED DESCRIPTION:
To clinically evaluate the treatment of mandibular class II furcation defects with enamel matrix derivative (EMD) and/or a bone substitute graft make of beta tricalcium phosphate/hydroxyapatite (βTCP/HA). Forty-one patients, presenting a mandibular class II buccal furcation defect, probing pocket depth (PPD) ≥ 4 mm and bleeding on probing, will be included. They will be randomly assigned to the groups: 1- EMD (n = 13); 2- βTCP/HA (n = 14); 3- EMD + βTCP/HA (n = 14). Relative gingival margin position (RGMP), relative vertical and horizontal attachment level (RVCAL and RHCAL) and PPD will be evaluated at baseline and 12 months. The mean horizontal clinical attachment level gain will be considered the primary outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, between 18-75 years of age;
* Presence of a mandibular molar with buccal class-II furcation defect, presenting PD ≥ 4mm, bleeding on probing (BOP), minimum (<1 mm) or no gingival recession after non-surgical therapy;
* Good general health;
* Minimum interproximal bone loss (< 2 mm).

Exclusion Criteria:

* Pregnant or lactating;
* Required antibiotic pre-medication for the performance of periodontal examination and treatment;
* Suffered from any other systemic diseases (cardiovascular, pulmonary, liver, cerebral, diseases or diabetes);
* Had received antibiotic treatment in the previous 3 months;
* Were taking long-term anti-inflammatory drugs;
* Had received a course of periodontal treatment within the last 6 months;
* Smokers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enilson A Sallum, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EMD + βTCP/HA: During flap access surgery, the granulation tissue will be removed and the root surfaces will be carefully instrumented with ultrasonic and hand instruments. The furcation will be filled with a mixture of enamel matrix derivative proteins (EMD) (Emdogain® Straumann, Basel, Switzerland) and bone substitute consisting of βTCP/HA (Bone Ceramic® Straumann, Basel, Switzerland). Immediately after debridement, EMD will be applied on the root surfaces.This mixture will be used to completely fill the defect (EMD + βTCP/HA).
Period: Overall Study
Arm/Group | EMD Alone | βTCP/HA Alone | EMD + βTCP/HA
Started | 13 | 14 | 14
Completed | 13 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Potential patients were selected from those referred to the Graduate Clinic of the Piracicaba Dental School. All patients received a complete periodontal examination, including anamnesis, a full-mouth periodontal probing, and radiographic examination. One furcation defect per patient was chosen, using Nabers probe.
Groups:
- Total: Total of all reporting groups
Arm/Group | βTCP/HA Alone | EMD + βTCP/HA | EMD Alone | Total
Number analyzed (Participants) | 14 | 14 | 13 | 41
Age, Customized [Count of Participants; unit: Participants] — Potential patients were selected from those referred to the Graduate Clinic of the Piracicaba Dental School. All patients received a complete periodontal examination, including anamnesis, a full-mouth periodontal probing, and radiographic examination.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 14 | 14 | 13 | 41
    >=65 years | 0 | 0 | 0 | 0
Age, Customized [Mean (Standard Deviation); unit: Years] | 53.69 (6.58) | 53.14 (5.92) | 54.57 (5.63) | 53.80 (5.92)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 10 | 8 | 27
  Male | 5 | 4 | 5 | 14
Plaque index (PI) [Mean (Standard Deviation); unit: Percent of surfaces with plaque] | 14.57 (3.83) | 14.36 (3.1) | 13.54 (2.99) | 14.17 (3.28)
Bleeding on probing (BOP) [Mean (Standard Deviation); unit: Percent of surfaces with bleeding] | 9.67 (3.1) | 9.68 (2.76) | 8.69 (1.84) | 9.36 (2.61)
Probing depth (PD) [Mean (Standard Deviation); unit: mm] | 4.92 (0.49) | 4.93 (0.73) | 4.79 (0.7) | 4.87 (0.64)
Relative gingival margin position (RGMP) [Mean (Standard Deviation); unit: mm] | 10.15 (0.9) | 9.57 (1.09) | 9.43 (1.34) | 9.60 (1.09)
Relative vertical clinical attachment level (RVCAL) [Mean (Standard Deviation); unit: mm] | 14.38 (1.76) | 14.64 (1.22) | 14.07 (1.44) | 14.36 (1.46)
Relative horizontal clinical attachment level (RHCAL) [Mean (Standard Deviation); unit: mm] | 5.08 (0.49) | 5.64 (0.93) | 5.5 (0.76) | 5.41 (0.77)

OUTCOME MEASURES:

1. Primary Outcome: Relative Horizontal Clinical Attachment Level (RHCAL) at 12 Months
Description: The relative horizontal clinical attachment level (RHCAL) will be measured with the same type of probe (PCP-15 Periodontal Probe - Hu-Friedy - Chicago, IL, USA) as the distance between the deepest point reached by the probe when introduced horizontally into the furcation and the lower border of the stent. This parameter will be evaluated at one specific site at the buccal furcation entrance, determined by a groove made on an individually manufactured acrylic stent and recorded to the nearest 0.5mm.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- βTCP/HA + EMD: During flap access surgery, the granulation tissue will be removed and the root surfaces will be carefully instrumented with ultrasonic and hand instruments. The furcation will be filled with a mixture of enamel matrix derivative proteins (EMD) (Emdogain® Straumann, Basel, Switzerland) and bone substitute consisting of βTCP/HA (Bone Ceramic® Straumann, Basel, Switzerland). Immediately after debridement, EMD will be applied on the root surfaces. The remaining part of the material in the seringe will be then mixed with the bone substitute on a sterile dappen. This mixture will be used to completely fill the defect (EMD + βTCP/HA).
  Flap access surgery: In the furcation sites, during flap access surgery, the granulation tissue will be removed and the root surfaces will be carefully instrumented with ultrasonic and hand instruments.
Arm/Group | βTCP/HA Alone | βTCP/HA + EMD | EMD Alone
Number analyzed (Participants) | 14 | 14 | 13
mm | 2.31 (0.75) | 3.00 (1.04) | 2.57 (0.94)

2. Secondary Outcome: Relative Vertical Clinical Attachment Level (RVCAL) at 12 Months
Description: The relative vertical clinical attachment level (RVCAL) will be measured with the same type of probe (PCP-15 Periodontal Probe - Hu-Friedy - Chicago, IL, USA) as the distance between the deepest point reached by the probe when introduced vertically into the buccal periodontal pocket. This parameter will be evaluated at one specific site at the buccal furcation entrance, determined by a groove made on an individually manufactured acrylic stent and recorded to the nearest 0.5mm.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | βTCP/HA Alone | EMD + βTCP/HA | EMD Alone
Number analyzed (Participants) | 14 | 14 | 13
mm | 12.31 (1.38) | 12.36 (1.5) | 11.93 (1.27)

3. Secondary Outcome: Periodontal Probing Depth at 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | EMD Alone | βTCP/HA Alone | EMD + βTCP/HA
Number analyzed (Participants) | 13 | 14 | 14
mm | 2.38 (0.65) | 2.57 (0.76) | 2.36 (1.08)

4. Secondary Outcome: Relative Gingival Margin Position (RGMP) at 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | EMD Alone | βTCP/HA Alone | EMD + βTCP/HA
Number analyzed (Participants) | 13 | 14 | 14
mm | 9.92 (1.12) | 9.79 (1.12) | 9.57 (1.02)

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Arm/Group | βTCP/HA Alone | βTCP/HA + EMD | EMD Alone
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This clinical trial did not show limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No